CLINICAL TRIAL: NCT03652948
Title: Evaluation of Meru Health Ascend Mobile Intervention for Depression in Middle Aged and Older Adults
Brief Title: Meru Health Ascend Mobile Intervention for Depression in Middle Aged and Older Adults
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: Meru Health, Inc. (Industry); Stanford University (Other)
Responsible Party: Principal Investigator, Christine Gould, Principal Investigator, Palo Alto Veterans Institute for Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOU0003
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Depression; Depressive Symptoms
Keywords: mobile app; middle age adults; older adults
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Study 1: 8 week mobile app based intervention using cognitive behavioral and mindfulness skills Study 2: 12 week mobile app based intervention (8 week intervention+4 weeks focused on sleep and nutrition)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meru Health Ascend Program (Experimental): The Meru Health Ascend Program is an 8-week mobile application (app) based intervention that teaches cognitive-behavioral and mindfulness skills. The intervention also includes a group discussion board with the other participants in the intervention group and therapist support via chat within the app.
  Study 2 is examining a revised version of the Meru Health Ascend Program that is 12 weeks long and incorporates sleep and nutrition information in addition to the 8-week program.
  Interventions: Behavioral: Meru Health Ascend Program

INTERVENTIONS:
Behavioral: Meru Health Ascend Program — Cognitive-behavioral skills, mindfulness

SUMMARY:
Using technology to deliver depression interventions is one way could alleviate the public health burden of depression. The study is testing a mobile app intervention program for depression that uses cognitive behavioral skills and mindfulness. This study seeks to obtain feedback on the intervention and refine the intervention and then test the intervention in a larger study. The mobile app intervention called the Meru Health Ascend program consists of the app and therapist support via messaging within the app.

DETAILED DESCRIPTION:
The Meru Health Ascend program is a guided self-management program that uses a mobile application to deliver content of the intervention. A licensed therapist (Meru Health employed) provides support to participants as needed and reviews practice logs within the app.The 8-week program teaches cognitive behavioral techniques and mindfulness skills with the aim of improving the user's mental health. The platform provides informational videos, skills practices, group discussion, and messaging with the therapist. The Meru Health program enrolls participants in treatment groups that work through the program at the same time and can provide support to on another on the discussion board within the app.

We are conducting two studies in middle aged and older adults with elevated depressive symptoms to evaluate the Meru Health Ascend program. In the first study (study 1), we will examine the feasibility of the intervention in individuals aged 40 years or older with elevated depression symptoms using an iterative case series. Specifically, we will examine the usability of app and materials, dropout and reasons for dropout, and user perceptions of the program.

We will then conduct a proof-of-concept study (study 2) using a nonrandomized pre-post design to examine whether individuals achieve clinically significant reductions in depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Owns a smart phone, resides in California, PHQ-9 score greater than or equal to 10, stable dose of medication (if taking psychotropic), able to read and understand English.

Exclusion Criteria:

* Psychotic disorder, possible cognitive impairment, evidence of problematic drinking behavior, active suicide ideation with a plan, active psychological treatment, bipolar disorder (study 2 only)

Ages: 40 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
change in depressive symptoms | Change from baseline to 8 weeks/posttreatment for study 1; change from baseline to 12 weeks for study 2
  The Patient Health Questionnaire 9-item (PHQ-9) is a measure that assesses 9 depressive symptoms with scores ranging from 0 to 27. Higher scores indicate more severe depressive symptomatology.

SECONDARY OUTCOMES:
change in anxiety symptoms | Change from baseline to 8 weeks/posttreatment for study 1; change from baseline to 12 weeks for study 2
  The Generalized Anxiety Disorder 7-item (GAD-7) is a seven item measure of anxiety symptoms with scores ranging from 0 to 21. Higher scores indicate more severe anxiety symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Gould, PhD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No